CLINICAL TRIAL: NCT01584830
Title: A Randomized, Double-blind, Placebo-controlled Phase III Study of Regorafenib Plus Best Supportive Care (BSC) Versus Placebo Plus BSC in Asian Subjects With Metastatic Colorectal Cancer (CRC) Who Have Progressed After Standard Therapy
Brief Title: Asian Subjects With Metastatic Colorectal Cancer Treated With Regorafenib or Placebo After Failure of Standard Therapy
Acronym: CONCUR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15808
Record Dates: First submitted 2012-04-24; First posted 2012-04-25 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-02

CONDITIONS: Colorectal Neoplasms
Keywords: Regorafenib; Colorectal; Metastatic
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — regorafenib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Regorafenib (BAY73-4506)
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Regorafenib (BAY73-4506) — Regorafenib BAY73-4506 will be given 3 weeks on/1 week off (160 mg od po.)
  Arms: Arm 1
Drug: Placebo — Placebo will be given 3 weeks on/1 week off (160 mg od po.)
  Arms: Arm 2

SUMMARY:
The purpose of this study is to assess if Regorafenib in combination with best supportive care will slow down tumor progression and result in increased survival in patients with metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological documentation of adenocarcinoma of the colon or rectum. All other histological types are excluded.
* Subjects with metastatic colorectal cancer(CRC) (Stage IV).
* Subjects must have failed at least two lines of prior treatment.
* Progression during or within 3 months following the last administration of approved standard therapies which must include a fluoropyrimidine, oxaliplatin and irinotecan.

  * Subjects treated with oxaliplatin in an adjuvant setting should have progressed during or within 6 months of completion of adjuvant therapy.
  * Subjects who progress more than 6 months after completion of oxaliplatin containing adjuvant treatment must be retreated with oxaliplatin-based therapy to be eligible.
  * Subjects who have withdrawn from standard treatment due to unacceptable toxicity warranting discontinuation of treatment and precluding retreatment with the same agent prior to progression of disease will also be allowed into the study.
  * Subjects may have received prior treatment with Avastin (bevacizumab) and/or Erbitux (cetuximab)/Vectibix (panitumumab) (if KRAS WT)
* Metastatic CRC subjects must have measurable or non measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria, version 1.1.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 1.
* Life expectancy of at least 3 months.
* Adequate bone marrow, liver and renal function as assessed by the laboratory required by protocol.

Exclusion Criteria:

* Prior treatment with Regorafenib.
* Previous or concurrent cancer that is distinct in primary site or histology from colorectal cancer within 5 years prior to randomization EXCEPT for curatively treated cervical cancer in situ, non-melanoma skin cancer and superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor invades lamina propria)].
* Extended field radiotherapy within 4 weeks or limited field radiotherapy within 2 weeks prior to randomization.
* Cardiological disease including Congestive heart failure, Unstable angina, Myocardial infarction, Cardiac arrhythmias requiring anti-arrhythmic therapy.
* Uncontrolled hypertension. (Systolic blood pressure 150 mmHg or diastolic pressure 90 mmHg despite optimal medical management).
* Subjects with phaeochromocytoma.
* Pleural effusion or ascites that causes respiratory compromise.
* Arterial or venous thrombotic or embolic events.
* Any history of or currently known brain metastases.
* Interstitial lung disease with ongoing signs and symptoms at the time of informed consent.
* Systemic anticancer therapy including cytotoxic therapy, signal transduction inhibitors, immunotherapy, and hormonal therapy during this trial or within 4 week.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2012-04; Primary Completion 2013-11 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | From randomization of the first subject untill 154 death events observed, up to 2 years
  OS is defined as the time from date of randomization to death due to any cause. Subjects still alive at the time of analysis were censored at their last date of last contact.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | From randomization of the first subject untill 154 death events observed, up to 2 years
  PFS was defined as the time from date of randomization to disease progression radiological/clinical or death due to any cause, whichever occurs first. Subjects without progression or death at the time of analysis were censored at their last date of tumor evaluation.
The percentage of subjects with total number of Complete Response (CR) + total number of Partial Response (PR). | From randomization of the first subject untill 154 death events observed, up to 2 years
Disease Control Rate (DCR) | From randomization of the first subject untill 154 death events observed, up to 2 years
  DCR is defined as the percentage of subjects whose best response was not Progressive Disease (PD) according to Response Evaluation Criteria in Solid Tumors (RECIST) (= total number of Complete Response (CR) + total number of Partial Response (PR) + total number of Stable Disease (SD); CR, PR, or SD had to be maintained for at least 28 days from the first demonstration of that rating)
Safety variables will be summarized using descriptive statistics based on adverse events collection | From randomization of the first subject untill 154 death events observed, up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (19):
- China (11):
  - Guangzhou, Guangdong
  - Harbin, Heilongjiang
  - Nanjing, Jiangsu
  - Xi'an, Shaanxi
  - Qingdao, Shandong
  - Chengdu, Sichuan
  - Hangzhou, Zhejiang
  - Beijing
  - Changchun
  - Shanghai
  - Tianjin
- Hong Kong (2):
  - Shatin, New Territories
  - Hong Kong
- Seoul, Korea, South Korea
- Taiwan (3):
  - Taipei, Taipei
  - Taipei
  - Taoyuan District
- Vietnam (2):
  - Hanoi
  - Ho Chi Minh City

REFERENCES:
- [Derived] Li J, Qin S, Xu R, Yau TC, Ma B, Pan H, Xu J, Bai Y, Chi Y, Wang L, Yeh KH, Bi F, Cheng Y, Le AT, Lin JK, Liu T, Ma D, Kappeler C, Kalmus J, Kim TW; CONCUR Investigators. Regorafenib plus best supportive care versus placebo plus best supportive care in Asian patients with previously treated metastatic colorectal cancer (CONCUR): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2015 Jun;16(6):619-29. doi: 10.1016/S1470-2045(15)70156-7. Epub 2015 May 13. PMID 25981818